CLINICAL TRIAL: NCT00063479
Title: Bisphosphonate Treatment of Osteogenesis Imperfecta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446H2202
Record Dates: First submitted 2003-06-27; First posted 2003-06-30 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; OI; bone markers; fracture; bone loss; pediatric; bisphosphonate; brittle bone disease; pamidronate
MeSH Terms: conditions — Osteogenesis Imperfecta; Fractures, Bone; Bone Diseases, Metabolic | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
The primary purpose of this trial is to evaluate whether the investigational medication is safe, effective and has the ability to increase spine bone density in osteogenesis imperfecta (OI) patients.

ELIGIBILITY:
Inclusion

* Male or Female children between 3 months and 17 years old
* OI type I, III or IV

Exclusion

* Deformity or abnormality which would prevent spine bone density from being done
* Any surgical bone-lengthening procedure
* Any kidney diseases or abnormalities
* Low calcium or vitamin D levels in the blood

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158
Dates: Start 2003-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in lumbar spine bone mineral density at month 12 relative to baseline

SECONDARY OUTCOMES:
Change in Z score of the lumbar spine at month 12 relative to baseline

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UCLA - Division of Pediatric Nephrology, Los Angeles, California
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Intermountain Orthopedics, Boise, Idaho
  - St. Jude Children's Research Hospital, Peoria, Illinois
  - Children's Hospital, Omaha, Nebraska
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hosptial, Houston, Texas